CLINICAL TRIAL: NCT02836808
Title: Validation of an Integrated Attention Model for Patients With Type 2 Diabetes
Acronym: CAIPADI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: dia-1190
Record Dates: First submitted 2016-04-08; First posted 2016-07-19 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2016-07

CONDITIONS: Type 2 Diabetes
Keywords: Multidisciplinary interventions; Long term control; Empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients attended with the standard model of care for diabetes, as out-patients in the Internal Medicine area
- CAIPaDi (Experimental): Patients attended in the Center of Comprehensive Care for the Patient with Diabetes, where they receive attention from 9 specialists in 1 day
  Interventions: Behavioral: CAIPaDi

INTERVENTIONS:
Behavioral: CAIPaDi — Patients are attended in 1 day by 9 specialists (endocrinologist, diabetes educators, nutritionist, psychologist, dentists, psychiatrist, physical activity specialist, foot care and ophthalmologist). They are attended in 4 monthly visits. After the initial phase, patients come back to the Center at 1 and 2 years for evaluation and reinforcement.
  Arms: CAIPaDi

SUMMARY:
Abstract: Empowerment interventions for chronic diseases are an evolving process. No agreement exists regarding the necessary components and methodologies to be applied. Systematic reviews have assessed the effect of self-management interventions. Improvements in illness beliefs, adherence to drug therapy and glucose monitoring have been reported. In the long term, no major changes have been achieved in weight, physical activity, smoking status, and depression scores.

There is a need for additional studies. The Center for Comprehensive Care of Patients with Diabetes (CAIPaDi) program is an intervention designed to provide education and empowerment techniques (using simple low-cost interactive tools) over a short period of time followed by at-distance support using internet or cell phone technology. The target population consists of patients with type 2 diabetes, free of chronic complications who are non-smokers. The intervention is composed of four monthly visits followed by a continuous at-distance support system. At each visit, patients stay for six hours in the center. Information is presented in group sessions. Empowerment techniques are applied during individual exchanges with the team or during facilitated group sessions. In summary, empowerment programs are an unmet need in many healthcare services.

DETAILED DESCRIPTION:
1. Background: There are major deficiencies in the attention quality provided to people with diabetes in Mexico. The percentage of compliance of therapeutic objectives is noticeably lower than the one informed in developed countries. It is required to have structured management strategies, adapted to traits of our population, which allow improving attention quality in the medium term. The National Institute of Medical Sciences and Nutrition Salvador Zubirán (INCMNSZ) developed an integrated management program by using the best evidence available. The target population is people with type 2 diabetes, with less than 5 years with the diagnosis, and is free from chronic complications. Selection criteria allow the intervention benefit to diminish incidence of chronic complications.
2. Hypothesis: "The management strategy applied at the Center of Comprehensive Care for the Patient with Diabetes (CAIPaDi) allows achieving the international treatment standards (proposed by NCQA) in a two-year period".
3. General and Specific objectives:

   General objective: To quantify the results one year after starting the integrated management program oriented to self-care activities applied at CAIPaDi.

   Specific objectives:
   * To measure the program impact (after 4 months, one and two years) based on the following variables: self-care (measured with standardized questionnaires), efficacy parameters (HbA1c, fasting glycemia, blood lipids, arterial pressure and use of anti-platelet aggregates), execution parameters (compliance of evaluations and preventive measures such as the search for microalbuminuria, ophthalmologic check, influenza vaccination, among others), incidence of micro- and macrovascular complications of diabetes, hospitalizations, use of emergency service or unforeseen expenses related to diabetes.
   * To compare the efficacy and execution parameters of the cases attended at the center, with patients with similar characteristics attended at the "Internal Medicine" service of the INCMNSZ.
   * To carry out a study of the social-economic impact of the intervention.
4. Goals: It is intended to validate an intervention that provides integrated attention to people with diabetes, in order to generate in the patient and his/her family, the competencies required for self-care in the long term and the prevention of chronic characteristics. Intervention is low-cost. This characteristic, along with the intervention systematization will allow the model to be exportable to the first-contact units.
5. Scientific Methodology: CAIPaDi has the mission of improving quality of life of patients with diabetes by means of an intervention adapted to the needs of patients, applying step-by-step action programs".

   Intervention consists of four monthly visits, each one being 6 hours long. The visits have individual and group sessions. The nine specialists in the multidisciplinary team are endocrinologists, diabetes educator, nutritionists, psychologist, dentists, psychiatrist, specialist in physical activity, ophthalmologist and foot care. Some of the functions may be fulfilled by the same health professional, previously trained.

   At each session, standardized actions are applied, which are assessed with preset indicators. At the initial and at yearly visits the following laboratory tests are taken: glycated hemoglobin, blood chemistry, lipid profile, liver function tests, albumin-creatinine index in an isolated urine sample, and 12-deviation electrocardiogram. At the yearly visits the patients receive reinforcement and treatment modifications as needed.

   Contact is kept with patients via phone calls, e-mails and messages on the mobile phone. Patients are asked to send their assessments on preset dates. Materials and tools are developed, which allow measuring information from the study in real time, empowerment of patients and decision-making by the multi-disciplinary team, based on clinical practice guidelines.

   There will be information from 1200 patients with 2-year follow-up. Besides having information from 1200 additional cases with follow-up at one year, and other 1200 others with assessments at 6 months. Therefore, the population for assessing execution variables shall be of 3600 participants. Such sample size allows us to detect differences higher than 5% in the percentage of cases that comply with the therapeutic objectives by comparing them with the initial assessment. As a secondary analysis, results will be compared with the population that receives attention the "Internal Medicine" service in the INCMNSZ (n=300 subjects).

   Patients will be referred from clinics or first contact physicians outside the Institute.
6. Expected impacts at medium and long term: This proposal allows validating the intervention designed and applied at CAIPaDi. In case of demonstrating its usefulness and cost-effectiveness, intervention will be exported to first-contact units. Manuals and tools have been developed which will allow the implementation of the program with minimum resources. Such action will allow creating a network of health units that operate with the same quality standards as INCMNSZ.
7. Infrastructure available at the participating institutions: The INCMNSZ has an area where the center operates.
8. Deliverable results: Procedure manuals for each of the actions included in the intervention, tools for decision making based on clinical practice guidelines which will be patented, educational materials designed for empowering patients (patentable products), an internet portal, an electronic file, a database, articles in high impact magazines, diploma courses for generating specific competencies related to diabetes treatment and to the center management.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 and under 70 years old
* having diagnosis of type 2 diabetes in the five previous years,
* having family support
* free of disabling diabetes complications

Exclusion Criteria:

* advanced complications of diabetes, such as ischemic heart disease, heart failure NYHA III-IV, KDOQI ≥3 renal failure, amputations, cerebral vascular disease, gastroparesis and muscular atrophy .
* type 1 diabetes mellitus, gestational diabetes or some variant of diabetes related to genetic syndromes, hyperlabile diabetes
* co-morbidities that limit their life expectancy such as malignant tumors
* advanced cognitive impairment or serious psychiatric disorders
* smoking, alcoholism or illegal drug dependence
* conditions that require surgical treatment in the short run or which prevent moderated activity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2013-10-31 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes control after 4 visits in a structured multidisciplinary program for patients with diabetes | 3 months
  HbA1c is measured in percentage (%). HbA1c will be compared from the first visit with the fourth visit.

SECONDARY OUTCOMES:
Diabetes control after 1 year in a structured multidisciplinary program for patients with diabetes | 1 year
  HbA1c is measured in percentage (%). HbA1c will be compared from the fourth visit with the visit 1 year apart.
Metabolic parameters are lipid profile after 1 year in a structured multidisciplinary program for patients with diabetes | 1 year
  Metabolic parameters are lipid profile (cholesterol, HDL cholesterol LDL cholesterol and triglycerides) in mg/dl. All of them will be compared from the fourth visit with the visit 1 year apart.
Renal function after 1 year in a structured multidisciplinary program for patients with diabetes | 1 year
  Renal function in mg/g (albumin/creatinine ratio). Renal function will be compared from the fourth visit with the visit 1 year apart.
Self-care by SDSCA questionnaire after 1 year in a structured multidisciplinary program for patients with diabetes | 1 year
  Self-care evaluation will be determined by SDSCA questionnaire and an objective examination of the patient doing the activities. This will be compared from the fourth visit with the visit 1 year apart.
Diabetic complications are eye, renal and foot evaluations after 1 year in a structured multidisciplinary program for patients with diabetes | 1 year
  Diabetic complications are eye, renal and foot evaluations. All of them will be compared from the fourth visit with the visit 1 year apart.
Quality of life after 1 year in a structured multidisciplinary program for patients with diabetes | 1 year
  Quality of life will be assessed with the DQoL (Diabetes Quality of Life) questionnaire. This will be compared from the fourth visit with the visit 1 year apart.
Diabetes control after 2 years in a structured multidisciplinary program for patients with diabetes | 2 years
  HbA1c is measured in percentage (%). HbA1c to be compared will be from fourth visit, 1 and 2 years apart.
Metabolic parameters are lipid profile after 2 years in a structured multidisciplinary program for patients with diabetes | 2 years
  Metabolic parameters are lipid profile (cholesterol, HDL cholesterol LDL cholesterol and triglycerides) in mg/dl. The parameters to be compared will be from fourth visit, 1 and 2 years apart.
Renal function after 2 years in a structured multidisciplinary program for patients with diabetes | 2 years
  Renal function in mg/g (albumin/creatinine ratio). The parameters to be compared will be from fourth visit, 1 and 2 years apart.
Self-care by SDSCA questionnaire after 2 years in a structured multidisciplinary program for patients with diabetes | 2 years
  Self-care evaluation will be determined by SDSCA questionnaire and an objective examination of the patient doing the activities. The parameters to be compared will be from fourth visit, 1 and 2 years apart.
Diabetic complications are eye, renal and foot after 2 years in a structured multidisciplinary program for patients with diabetes | 2 years
  Diabetic complications are eye, renal and foot evaluations. All of them will be compared from the fourth visit with the visit 1 year apart. The parameters to be compared will be from fourth visit, 1 and 2 years apart.
Quality of life after 2 years in a structured multidisciplinary program for patients with diabetes | 2 years
  Quality of life will be assessed with the DQoL (Diabetes Quality of Life) questionnaire. The parameters to be compared will be from fourth visit, 1 and 2 years apart.
Metabolic parameters are lipid profile after 4 visits in a structured multidisciplinary program for patients with diabetes | 3 months
  Metabolic parameters are lipid profile (cholesterol, HDL cholesterol LDL cholesterol and triglycerides) in mg/dl. All of them will be compared from the first visit with the fourth visit.
Renal function after 4 visits in a structured multidisciplinary program for patients with diabetes | 3 months
  Renal function in mg/g (albumin/creatinine ratio). Renal function will be compared from the first visit with the fourth visit.
Self-care by SDSCA questionnaire after 4 visits in a structured multidisciplinary program for patients with diabetes | 3 months
  Self-care evaluation will be determined by SDSCA questionnaire and an objective.
Diabetic complications are eye, renal and foot evaluations after 4 visits in a structured multidisciplinary program for patients with diabetes | 3 months
  Diabetic complications are eye, renal and foot evaluations. All of them will be compared from the first visit with the fourth visit.
Quality of life after 4 visits in a structured multidisciplinary program for patients with diabetes | 3 months
  Quality of life will be assessed with the DQoL (Diabetes Quality of Life) questionnaire. This will be compared from the first visit with the fourth visit.

OTHER OUTCOMES:
Glucose control of the cases attended at the Center compared with those of patients with similar characteristics attended in the "Internal Medicine" service of the INCMNSZ. | 2 years
  HbA1c is measured in percentage (%). Comparison will be with patients from the Internal Medicine ward, who meet the same clinical characteristics as the patients from the Center.
Lipid parameters of the cases attended at the Center compared with those of patients with similar characteristics attended in the "Internal Medicine" service of the INCMNSZ. | 2 years
  Metabolic parameters are lipid profile (cholesterol, HDL cholesterol LDL cholesterol and triglycerides) in mg/dl. Comparison will be with patients from the Internal Medicine ward, who meet the same clinical characteristics as the patients from the Center.
Renal function evaluation of the cases attended at the Center compared with those of patients with similar characteristics attended in the "Internal Medicine" service of the INCMNSZ. | 2 years
  Renal function in mg/g (albumin/creatinine ratio). Comparison will be with patients from the Internal Medicine ward, who meet the same clinical characteristics as the patients from the Center.
Self-care evaluation of the cases attended at the Center compared with those of patients with similar characteristics attended in the "Internal Medicine" service of the INCMNSZ. | 2 years
  Self-care evaluation will be determined by SDSCA questionnaire and an objective examination of the patient doing the activities. Comparison will be with patients from the Internal Medicine ward, who meet the same clinical characteristics as the patients from the Center.
Evaluation of complications of the cases attended at the Center compared with those of patients with similar characteristics attended in the "Internal Medicine" service of the INCMNSZ. | 2 years
  Diabetic complications are eye, renal and foot evaluations. Comparison will be with patients from the Internal Medicine ward, who meet the same clinical characteristics as the patients from the Center.
Quality of life of the cases attended at the Center compared with those of patients with similar characteristics attended in the "Internal Medicine" service of the INCMNSZ. | 2 years
  Quality of life will be assessed with the DQoL (Diabetes Quality of Life) questionnaire. Comparison will be with patients from the Internal Medicine ward, who meet the same clinical characteristics as the patients from the Center.
Social-economic impact of expenses on food of a multidisciplinary intervention for patients with diabetes | 2 years
  Patients will be asked about expenses on food. It will be included an evaluation of visits to emergency service related to diabetes complications and costs generated from this visit.
Social-economic impact of exercising facilities and usage of a multidisciplinary intervention for patients with diabetes | 2 years
  Patients will be asked about the expense for the use of facilities for exercise at the beginning and at the fourth visit.
Social-economic impact of drug treatment of a multidisciplinary intervention for patients with diabetes | 2 years
  Patients will be asked about the expense drug treatment at the beginning and at the fourth visit. It will be included an evaluation of visits to emergency service related to diabetes complications and costs generated from this visit.
Social-economic impact of transportation of a multidisciplinary intervention for patients with diabetes | 2 years
  Patients will be asked about the expense transportation at the beginning and at the fourth visit. It will be included an evaluation of visits to emergency service related to diabetes complications and costs generated from this visit.
Social-economic impact of living and eating expenses of a multidisciplinary intervention for patients with diabetes | 2 years
  Patients will be asked about the expense living and eating at the beginning and at the fourth visit. It will be included an evaluation of visits to emergency service related to diabetes complications and costs generated from this visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio C Hernández, MD, Principal Investigator — National Institute of Medical Sciences and Nutrition Salvador Zubirán
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Journal publication. The information to be shared will be metabolic parameters and questionaire results. The data will be available on 2016. Metabolic parameters will be obtained from blood samples and the questionnaires results from those self-applied or applied during praxis.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: January 2018. The data will be available for 5 years
Access Criteria: Undefined

REFERENCES:
- [Background] Villalpando S, Shamah-Levy T, Rojas R, Aguilar-Salinas CA. Trends for type 2 diabetes and other cardiovascular risk factors in Mexico from 1993-2006. Salud Publica Mex. 2010;52 Suppl 1:S72-9. doi: 10.1590/s0036-36342010000700011. PMID 20585732
- [Background] Aguilar Salinas CA, Gómez Diaz RA, Gomez Perez FJ. Diabetes en Mexico: Principales retos y posibles soluciones. Revista ALAD 2011: 19:146-161
- [Background] Tricco AC, Ivers NM, Grimshaw JM, Moher D, Turner L, Galipeau J, Halperin I, Vachon B, Ramsay T, Manns B, Tonelli M, Shojania K. Effectiveness of quality improvement strategies on the management of diabetes: a systematic review and meta-analysis. Lancet. 2012 Jun 16;379(9833):2252-61. doi: 10.1016/S0140-6736(12)60480-2. Epub 2012 Jun 9. PMID 22683130
- [Background] Planas LG, Crosby KM, Farmer KC, Harrison DL. Evaluation of a diabetes management program using selected HEDIS measures. J Am Pharm Assoc (2003). 2012;52(6):e130-8. doi: 10.1331/JAPhA.2012.11148. PMID 23224336
- [Background] Hernandez-Jimenez S, Garcia-Ulloa C, Mehta R, Aguilar-Salinas CA, Kershenobich-Stalnikowitz D. Innovative models for the empowerment of patients with type 2 diabetes: the CAIPaDi program. Recent Pat Endocr Metab Immune Drug Discov. 2014;8(3):202-9. doi: 10.2174/1872214808999141110155515. PMID 25381833
- [Derived] Landa-Anell MV, Del Razo-Olvera FM, Bodnar I, Cordova-Isidro B, Lagunas-Valdepena D, Arias-Marroquin AT, Garcia-Ulloa AC, Melgarejo-Hernandez MA, Hernandez-Jimenez S; Group of Study CAIPaDi. Nutritional diagnoses in people with type 2 diabetes: association with metabolic, anthropometric, and dietary parameters. Front Nutr. 2024 Oct 18;11:1473429. doi: 10.3389/fnut.2024.1473429. eCollection 2024. PMID 39494309
- [Derived] Garcia-Ulloa AC, Almeda-Valdes P, Cuatecontzi-Xochitiotzi TE, Ramirez-Garcia JA, Diaz-Pineda M, Garnica-Carrillo F, Gonzalez-Duarte A, Narayan KMV, Aguilar-Salinas CA, Hernandez-Jimenez S; CAIPaDi Study Group. Detection of sudomotor alterations evaluated by Sudoscan in patients with recently diagnosed type 2 diabetes. BMJ Open Diabetes Res Care. 2022 Dec;10(6):e003005. doi: 10.1136/bmjdrc-2022-003005. PMID 36521878
- [Derived] Garcia-Ulloa AC, Lechuga-Fonseca C, Del Razo-Olvera FM, Aguilar-Salinas CA, Galaviz KI, Narayan KMV, Hernandez-Jimenez S; Group of Study CAIPaDi. Clinician prescription of lipid-lowering drugs and achievement of treatment goals in patients with newly diagnosed type 2 diabetes mellitus. BMJ Open Diabetes Res Care. 2021 Feb;9(1):e001891. doi: 10.1136/bmjdrc-2020-001891. PMID 33568360